CLINICAL TRIAL: NCT01880593
Title: Ketamine Plus Lithium as a Novel Pharmacotherapeutic Strategy in Treatment-Resistant Depression
Brief Title: Ketamine Plus Lithium in Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 13-0365
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Depression
Keywords: Ketamine; glutamate; N-methyl-D-aspartate; depression; major depressive disorder; treatment resistant; antidepressant; lithium
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Lithium; Lithium Carbonate; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine and Lithium (Experimental): Subjects in this arm take 600-1200mg of Lithium pills at night for duration of the study
  Interventions: Drug: Lithium; Drug: Ketamine
- Ketamine and Placebo (Placebo Comparator): Subjects in this arm take placebo pills at night for duration of the study.
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Subjects in this arm take 600-1200mg of Lithium pills at night for duration of the study.
  Other Names: Lithium Carbonate Immediate Release
  Arms: Ketamine and Lithium
Drug: Ketamine
Drug: Placebo — Subjects in this arm take placebo pills at night for duration of the study.
  Arms: Ketamine and Placebo

SUMMARY:
The purpose of this study is to test the antidepressant effect of ketamine when given repeatedly over a period of 1 week, as well as the use of Lithium as a relapse-prevention strategy for patients with treatment-resistant depression (TRD) who respond to an initial series of ketamine infusions. Ketamine is a Food and Drug Administration approved anesthetic (a drug used to produce loss of consciousness before and during surgery). Ketamine is not approved for the treatment of major depressive disorder and is considered experimental in this study. An additional purpose of this study is to research the effects of ketamine on brain function.

You may qualify to take part in this research study because you have been diagnosed with major depressive disorder (MDD) and have not responded to past treatments.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a disabling medical illness and current monoaminergic treatments are slow to act and possess only limited efficacy. In this context, the discovery that the glutamate NMDA receptor antagonist ketamine is rapidly antidepressant (onset of action within hours) -- even in patients suffering from treatment-resistant depression (TRD) -- has ignited tremendous enthusiasm among clinicians, scientists and patients alike. A critical obstacle to the translation of this discovery into a novel treatment, however, is the limited duration of action following a course of ketamine (e.g. 1-2 weeks). The current project will address this important gap in medical knowledge by testing a rational neuropharmacological strategy designed to optimize and sustain the rapid antidepressant effects of ketamine. Driven by the recent characterization of the molecular mechanisms underpinning the antidepressant and neuroplasticity effects of ketamine, we will test the combination of ketamine plus lithium in patients with TRD using a randomized, double blind, placebo-controlled design. The primary aims of the project are (1) to test the efficacy of lithium-plus-ketamine compared to placebo-plus-ketamine as an antidepressant combination strategy in TRD and (2) to gather data on the safety and tolerability of the lithium-plus-ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 21-65 years of age;
* Female individuals who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or using a medically accepted reliable means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative serum B-HCG at screening and at pre-infusion;
* Participants must fulfill DSM-IV criteria for Major Depression without psychotic features, based on clinical assessment by a study psychiatrist and confirmed by a structured diagnostic interview, the Structured Clinical Interview for DSM-IV TR Axis I Disorders, Patient Edition (SCID-P);
* Participants must have a history of at least one previous episode of depression prior to the current episode (recurrent MDD) or have chronic MDD (of at least two years' duration);
* Participants have not responded to two or more adequate trials of an antidepressant as determined by Antidepressant Treatment History Form (ATHF) criteria (score >=3);
* Current Major Depressive Episode of at least moderate severity, defined as a QIDS-SR score ≥ 14 and a CGI-S score of ≥ 4;Current major depressive episode is of at least 4 weeks duration;
* Each participant must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document;
* Each participant must be able to identify a family member, physician, or friend who will participate in the Treatment Contract.

Exclusion Criteria:

* Lifetime history of psychotic features, diagnosis of schizophrenia or any other psychotic disorder, or diagnosis of bipolar disorder;
* Lifetime histories of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
* Current diagnosis of OCD or eating disorder (bulimia nervosa or anorexia nervosa);
* Subjects with DSM-IV drug or alcohol abuse/dependence within the preceding 2 years;
* Patients with schizotypal or antisocial personality disorder, or any clinically significant axis II disorder that would, in the investigator's judgment, preclude safe study participation;
* Patients judged clinically to be at serious and imminent suicidal or homicidal risk;
* Women who are either pregnant or nursing;
* Serious, unstable medical illnesses including hepatic, renal impairment, gastroenterologic (including gastro-esophageal reflux disease), respiratory (including obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics), cardiovascular (including ischemic heart disease and uncontrolled hypertension), endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
* Patients who have a positive urine toxicology for illicit substances at screening and within 24 hours of the infusion;
* Patients with one or more seizures without a clear and resolved etiology;
* Treatment with an irreversible MAOI within 2 weeks prior to randomization or fluoxetine within 4 weeks prior to randomization;
* Treatment with other antidepressants within one week of randomization;
* Previous recreational use of PCP or ketamine;
* Hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg) not controlled by diuretic or beta-blocker therapy alone or in combination;
* A blood pressure reading over 160/90 or two separate readings over 140/90 at screening or baseline visits;
* Renal impairment, as reflected by a BUN > 20 mg/dL and/or creatinin clearance of >1.3 mg/dL;
* Thyroid impairment, as reflected by a TSH > 4.2 mU/L;
* Cardiac disease, as reflected by an EKG that is abnormal and of concern for cardiac disease;
* Any anticipated change in medications that could affect fluid or salt balance, including the following antihypertensive agents: ACE inhibitor, loop diuretics, calcium channel blockers, thiazide diuretics, angiotensin II receptor blockers.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from May 2013 through Sept 2016
Groups:
- Ketamine and Lithium: 600-1200mg of Lithium pills at night for duration of the study
- Ketamine and Placebo: Placebo pills at night for duration of the study
Period: Overall Study
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Started | 18 | 16
Completed | 10 | 10
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 5
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine and Lithium | Ketamine and Placebo | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12.65) | 45.87 (10.94) | 45.41 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 7 | 16
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
  units on a scale | 32.39 (3.87) | 32.81 (5.61) | 32.58 (4.69)
QIDS [Mean (Standard Deviation); unit: units on a scale] — Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) score - Each item is rated 0 to 3. The total score ranges from 0 (no depression) - 27 (severe depression).
  units on a scale | 16.22 (4.33) | 18.19 (3.082) | 17.16 (4.32)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 4.66 (.59) | 5 (.52) | 4.92 (.57)
BSS [Mean (Standard Deviation); unit: units on a scale] — BECK Scale for Suicidal Ideation (BSS) - 0-13 Minimal; 14-19 Mild; 20-28 Moderate; 29-63 Severe
  units on a scale | 5.89 (7.71) | 7.56 (8.31) | 7.24 (8.10)
HAM-A [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Rating Scale (HAM-A). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
  units on a scale | 18.78 (7.02) | 20.31 (5.11) | 19.5 (6.15)
CSSRS (lifetime) [Mean (Standard Deviation); unit: units on a scale] — The Columbia-Suicide Severity Rating Scale (C-SSRS) - Full range from 0 (low intensity suicidal ideation to 9 (high intensity suicidal ideation).
  units on a scale | 2.5 (2.7) | 2.06 (2.02) | 2.29 (2.28)

OUTCOME MEASURES:

1. Primary Outcome: MADRS-S Score
Description: The Montgomery Asberg Depression Rating Scale (MADRS-S) has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Time Frame: 2 weeks after last ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 22.56 (11.22) | 23 (12.6)

2. Secondary Outcome: QIDS-SR Score
Description: Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) score - Each item is rated 0 (no depression) to 3 (severe depression), for a total score range of 0 (no depression) to 27 (severe depression).
Time Frame: 2 weeks after last ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 9.89 (6.04) | 10.13 (6.47)

3. Secondary Outcome: CGI-S Score
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: 2 weeks after last ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 3.83 (.86) | 3.875 (1.36)

4. Secondary Outcome: HAM-A Score
Description: Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: 2 weeks after last ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 13.5 (8.15) | 11.13 (6.08)

5. Secondary Outcome: BSS Score
Description: BECK Scale for Suicidal Ideation (BSS) - 0-13 Minimal; 14-19 Mild; 20-28 Moderate; 29-63 Severe
Time Frame: 2 weeks after last ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 4.94 (7.35) | 2.69 (5.95)

6. Secondary Outcome: CSSRS Score
Description: Columbia Suicide Severity Rating Scale (CSSRS) - Full range from 0 (low intensity suicidal ideation to 9 (high intensity suicidal ideation).
Time Frame: 2 weeks after last ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | .833 (2.12) | .44 (.89)

7. Secondary Outcome: Patient Rated Inventory of Side Effects (PRISE)
Description: Number of Participants with PRISE
Time Frame: 2 weeks after last ketamine infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
Number analyzed (Participants) | 18 | 16
Participants | 3 | 2

ADVERSE EVENTS:
Arm/Group | Ketamine and Lithium | Ketamine and Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 15/18 | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine and Lithium (N=18) | Ketamine and Placebo (N=16)
Nausea (Gastrointestinal disorders) | 8 | 4
Dry Mouth (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 9 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 8 | 9
Dizziness (Nervous system disorders) | 2 | 0
Tinnitus (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Chest Discomfort (General disorders) | 0 | 2
Pollakiuria (Renal and urinary disorders) | 3 | 1
Polyuria (Renal and urinary disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes